CLINICAL TRIAL: NCT07262645
Title: A Multicenter, Randomized, Double-Blind, Sham-Controlled Study on The Efficacy And Safety of Near-Infrared Light Therapy Device in Participants With Mild-Moderate Alzheimer's Disease (NirsCure-03A)
Brief Title: Near-infrared Light Therapy Device for Mild-Moderate Alzheimer's Disease (NirsCure-03A)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Danyang Huichuang Medical Equipment Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NirsCure-03A
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer s Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham device (Sham Comparator): Device: NirsCure 6000 sham device (once daily for 30 minutes, six times per week)
  Interventions: Device: Sham Device
- Near infrared light therapy (Experimental): Device: NirsCure 6000 Near-infrared light therapy (once daily for 30 minutes, six times per week)
  Interventions: Device: NirsCure 6000

INTERVENTIONS:
Device: NirsCure 6000 — Near-infrared light therapy. Once daily for 30 minutes, six times per week.
  Arms: Near infrared light therapy
Device: Sham Device — Sham device (once daily for 30 minutes, six times per week)
  Arms: Sham device

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo (sham device)-controlled clinical trial.

A total of 320 patients with mild to moderate Alzheimer's disease (AD) are planned to be enrolled. Central stratified block randomization will be applied, with stratification based on disease severity (mild vs. moderate) and PET subgroup participation status (yes vs. no). Participants will be randomly assigned to either the treatment group or control group in a 1:1 ratio. After enrollment, participants will complete the treatment at home. The treatment group will receive therapy using a near-infrared light therapy device, while the control group will use sham device. Both investigators and participants will remain blinded to treatment allocation throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged between 50 to 85 years old (inclusive).
2. Participants must have at least 4 years of formal education and be capable of completing cognitive and other protocol-specified assessments.
3. Documented progressive memory decline for ≥12 months prior to screening.
4. Meets the core clinical diagnostic criteria for mild to moderate AD dementia (stages 4-5), according to the National Institute on Aging and the Alzheimer's Association (NIA-AA) 2018 research framework and the AA workgroup 2024 update.
5. Evidence of positive brain amyloid pathology, demonstrated by at least one of the following:

   1. Positive Aβ-PET scan (historical positive result acceptable); or
   2. Positive Cerebrospinal fluid (CSF) Aβ testing (historical positive result acceptable).
6. Mini-Mental State Examination (MMSE) total score between 15 and 26 inclusive (between 12 and 22 for participants with an elementary school education level).
7. Clinical Dementia Rating (CDR) Global of 1 or 2, and the CDR-Memory Box scores ≥ 0.5.
8. If receiving acetylcholinesterase inhibitor or memantine, participants must be on a stable dose for at least 12 weeks prior to baseline.
9. Must have at least one reliable study partner who can accompany the participant to complete daily treatment. The study partner should have a close relationship with the participant and sufficient knowledge to accurately report on cognition, function, behavior, safety, and protocol compliance. The study partner must be able to communicate with study staff via phone or WeChat, attend required on-site visit, provide informed consent to supporting follow-up throughout the study.
10. The participant, study partner, or legally authorized representative voluntarily agrees to participate and provides written informed consent prior to any study procedures.

Exclusion Criteria:

1. Presence of any diagnosis other than AD that could cause dementia or cognitive decline, including but not limited to: vascular dementia; Central nervous system infections (e.g., HIV, neurosyphilis); Creutzfeldt-Jakob disease; Huntington's disease; Parkinson's disease; Lewy body dementia; Traumatic brain injury-related dementia; Dementia caused by physical and chemical factors (e.g., drug toxicity, alcohol intoxication, carbon monoxide poisoning); significant systemic diseases (e.g., hepatic or pulmonary encephalopathy); Intracranial space-occupying lesions (e.g., subdural hematoma, brain tumors); or dementia clearly attributable to endocrine disorders, vitamin deficiencies, or other identifiable causes.
2. Brain MRI demonstrating significant pathological findings, including but not limited to:

   1. More than two infarcts with a diameter > 2 cm, or a single infarct involving critical regions (thalamus, hippocampus, entorhinal cortex, parahippocampal cortex, angular gyrus, or other cortical and subcortical gray matter nuclei);
   2. Extensive white matter hyperintensities (Fazekas score ≥ 3);
   3. Space-occupying lesions such as cysts, abscesses, or brain tumors (e.g., meningiomas or arachnoid cysts). Specifically, meningiomas or arachnoid cysts with a maximum diameter < 1 cm do not require exclusion.
3. History of transient ischemic attack (TIA), stroke, or seizure within 6 months of screening.
4. Hachinski Ischemic Score (HIS) > 4.
5. Hamilton Depression Rating Scale (HAMD-17) total score > 10.
6. Diagnosis of a psychiatric disorder according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) at screening, including schizophrenia or other psychotic disorders, bipolar disorder, major depressive disorder, or delirium.
7. Known history or laboratory confirmation of HIV infection or neurosyphilis at screening.
8. Severe cardiovascular disease, including New York Heart Association (NYHA) class III or IV heart function; Severe or unstable angina, or newly developed unstable angina within 3 months prior to screening (with objective clinical evidence such as cardiac enzyme abnormalities or dynamic ST-T changes on electrocardiogram); Acute myocardial infarction within 6 months prior to screening.
9. Severe dysfunction of major organs (heart, lungs, liver, kidneys, etc.), or any medical condition that, in the opinion of the investigator, could render the participant unsuitable for this study or interfere with participation.
10. Current or prior treatment with any anti-amyloid monoclonal antibody (e.g., aducanumab, lecanemab, or donanemab).
11. Prior or planned lymphaticovenous anastomosis (LVA) of the cervical deep lymphatic vessels.
12. Participation in any interventional clinical trial involving a drug or medical device within the 30 days prior to screening, except for observational studies or verified placebo-group participation in a previous interventional trial.
13. History of severe head trauma or implanted cranial devices (e.g., bone screws, bone plates, prior cranial surgery, deep brain stimulators); Contraindications to MRI (e.g., claustrophobia, pacemakers/defibrillators, ferromagnetic metal implants); unwilling to undergo MRI examination.
14. Contraindications to PET or allergy to Aβ-PET tracer (except participants enrolled based solely on CSF Aβ positivity). Participants with uncontrolled abnormal blood glucose, allergy to FDG tracer, or any other investigator-judged contraindications are ineligible for the FDG-PET substudy.
15. History of malignancy within 5 years prior to screening, except for:

    1. Adequately treated basal or squamous cell skin carcinoma, or cervical dysplasia;
    2. Adequately treated Stage I in situ cervical cancer ≥ 2 years prior to screening without recurrence;
    3. Prostate cancer confined to the prostate, adequately treated (e.g., surgery, radiotherapy, or active surveillance), with stable prostate-specific antigen (PSA) levels for ≥ 2 years prior to screening;
    4. Non-metastatic breast cancer, adequately treated and without recurrence.
16. Women who are pregnant, breastfeeding, planning pregnancy, or of childbearing potential not using highly effective contraception.
17. Any other condition that, in the opinion of the investigator, may compromise the participant's safety, interfere with protocol adherence, or confound study results.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 320 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-07-22 (Estimated); Study Completion 2027-07-22 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale, cognitive subscale 13 (ADAS-Cog13) | 26 weeks
  Change from baseline in Alzheimer's Disease Assessment Scale - Cognitive Subscale 13 (ADAS-Cog13) score at 26-Weeks. The ADAS-Cog13 score ranges from 0 to 85, with higher scores indicating greater cognitive impairment.

SECONDARY OUTCOMES:
Clinical Dementia Rating - Sum of Boxes (CDR-SB) | 26 weeks
  Change from baseline in Clinical Dementia Rating - Sum of Boxes (CDR-SB) score at 26-Weeks. The CDR-SB score ranges from 0 to 18, with higher scores indicating greater cognitive and functional impairment.
Mini-Mental Status Examination (MMSE) | 26 weeks
  Change from baseline in Mini-Mental State Examination (MMSE) score at 26-Weeks. The MMSE score ranges from 0 to 30, with higher scores indicating better cognitive function.
Alzheimer's Disease Cooperative Study Activities of Daily Living Scale (ADCS-ADL) | 26 weeks
  Change from baseline in Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL) score at 26-Weeks. The ADCS-ADL score ranges from 0 to 78, with higher scores indicating better functional ability in activities of daily living.
Integrated Alzheimer's Disease Rating Scale (iADRS) | 26 weeks
  Change from baseline in Integrated Alzheimer's Disease Rating Scale (iADRS) score at 26-Weeks. The iADRS score ranges from 0 to 144, with higher scores indicating better overall cognitive and functional performance.

CONTACTS AND LOCATIONS:
Locations (23):
- China (23):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Shijiazhuang People's Hospital, Shijiazhuang, Hebei
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Tangdu Hospital, Air Force Medical University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Pudong Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - General Hospital, Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Huanhu Hospital, Tianjin, Tianjin Municipality
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang